CLINICAL TRIAL: NCT05886309
Title: Measurement of Serum Ferritin With a Cryo Detector Mass Spectrometer (CDMS): Pilot Study and First Experience in Testing Human Serum
Brief Title: Measurement of Serum Ferritin With a Cryo Detector Mass Spectrometer (CDMS)
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Metromol SA (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-00550; th22Infanti
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Serum Ferritin
Keywords: Cryo Detector Mass Spectrometer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Collection of Blood samples — The following samples will be drawn from each study participant immediately after the venipuncture performed for the whole blood donation:
  * 1 sample with no anticoagulant (5 ml) for SF measurement with the CDMS method
  * 1 EDTA (Ethylendiamintetraazetat) sample (7,5 ml) for a complete blood count with red blood cell indices and reticulocytes
  * 1 EDTA sample (2,7 ml) for the measurement of hepcidin
  * 1 Li-Heparin-Gel sample (4.7 ml) for the measurement of SF with the ECLIA (Electrochemiluminescence-enzymeimmunoassay) and of the complete set of iron biomarkers (Transferrin Saturation, serum iron, Soluble Transferrin Receptor)
  * 1 Li-Heparin-Gel sample (4.7 ml) for the measurement of CRP (C-reactive Protein)
  * 1 sample with no anticoagulant (5 ml) for the measurement of SF with the CMIA (Chemiluminescence Immunoassay)
  * 1 sample with no anticoagulant (5 ml) for storage

SUMMARY:
The study will explore the performance of the CDMS (Cryo Detector Mass Spectrometer) method in measuring SF (serum ferritin) in human serum of healthy individuals. This will be the first experience of testing SF with this method using biologic material of human origin.

DETAILED DESCRIPTION:
A clear interpretation of hyperferritinemia is difficult in many clinical situations. Crucial for the correct treatment of patients is the differentiation between reactively elevated ferritin and effective iron overload.The measurement methods that are routinely used provide quantitative results of the measurement of total ferritin molecules independent of their actual iron content.With a modified mass spectrometric method (CDMS), this should be possible.

In this study the investigators would like to apply this measurement technique for the first time with human serum as the investigators would like to test healthy blood donors with known normal, low or elevated ferritin levels.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* SF (serum ferritin) values known from a previous determination that must not be older than twelve months and not followed by a blood donation
* fulfillment of the eligibility criteria for blood donation
* negative serology for HBV (hepatitis B virus), HCV (hepatitis C virus), HIV (human immunodeficiency virus) as assessed in the context of a blood donation

Exclusion Criteria:

* acute illness
* chronic inflammatory disease

Since pregnancy is a contraindication for blood donation, no pregnant women will be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study cohort will include 20-25 experienced blood donors (not first-time donors) distributed among three groups according to SF values obtained from at least two previous measurements:
  * low SF levels: < 20 ng/ml
  * normal SF levels: 50-200 ng/ml (women) or 50-300 ng/ml (men)
  * high SF levels: > 200 ng/ml (women) or > 300 ng/ml (men)
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Assessment of the mass of serum ferritin molecules (kDa) | one time assessment at baseline
  The primary outcome is the mass of SF molecules measured using the CDMS method

CONTACTS AND LOCATIONS:
Overall Officials: Laura Infanti, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland